CLINICAL TRIAL: NCT00105365
Title: Shoe Modification and Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3120-P
Record Dates: First submitted 2005-03-11; First posted 2005-03-14 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Knee Osteoarthritis
Keywords: lateral wedge inserts; shoe inserts
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- walking shoes (Placebo Comparator): walking shoes
  Interventions: Other: walking shoes
- walking shoes + shoe insert (Experimental): walking shoes + shoe insert
  Interventions: Device: Shoe insert

INTERVENTIONS:
Device: Shoe insert — Subjects with knee OA underwent gait analysis and knee pain and function assessment at baseline while wearing walking shoes and after four weeks of wearing walking shoes with lateral-wedged insoles.
  Arms: walking shoes + shoe insert
Other: walking shoes — walking shoes
  Arms: walking shoes

SUMMARY:
This trial will assess the ability of shoe inserts to relieve pain and disability in people with knee osteoarthritis (OA) in the inner (medial) aspect of the knee.

DETAILED DESCRIPTION:
Osteoarthritis (OA), the most common joint disease in humans, is a significant cause of pain and disability. Its prevalence increases with age, leading to about 65-85% of those age 65 years and older having OA. Involvement of the knee with OA is the main reason for significant functional impairment as it alters ambulation through pain and stiffness. Nonpharmacological management of knee OA includes the use of orthotic supports such as wedged insoles for varus or valgus knee deformities to relieve pain and improve function in the early stages of this joint disease. Although these interventions are desirable because they are simple and inexpensive, we do not have a clear understanding about their efficacy in relieving pain and disability in people with knee OA. We also do not know whether there is a relationship between changes in joint biomechanics that occur with wedged insoles and changes in function and progression of OA. Furthermore, information is lacking regarding which patients would benefit from wedged insoles. Answering these questions will be critically important in the development of guidelines for the prescription of wedged insoles in knee OA. Patients in this study will be evaluated at baseline and after wearing the lateral-wedged insoles immediately and after wearing the insoles for four weeks. The participants will wear lateral-wedged insoles for the painful knee(s) for as many hours and for as many days of the week as they can tolerate. Some subjects may use a neutral position insole for an asymptomatic knee.

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk 30 feet without a walking aid
* Ability to stand unaided
* Ability to understand verbal instructions
* Ability to give informed consent

Exclusion Criteria:

* History of knee trauma or surgery including arthroscopic surgery in the past 6 months
* Severe obesity (>30 kg/m2)
* Neurological disease
* Injury or amputation to the lower extremity joints
* History of other types of arthritis
* Symptomatic spine, hip, ankle, or foot disease that would interfere with assessment of the knee
* Intra-articular steroids in the past 3 months, or hyaluronic acid in the last 6 months
* Poor health that would impair compliance or assessment such as shortness of breath with exertion

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-03; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
WOMAC pain scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Meika A Fang, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States